CLINICAL TRIAL: NCT05935917
Title: A Phase 1, Open-label, Single-dose, Randomized, Two-period, Crossover Study Evaluating the Bioequivalence of Brincidofovir Form H and Form II Tablets in Healthy Adult Participants
Brief Title: Study Evaluating the Bioequivalence of Brincidofovir Form H and Form II Tablets in Healthy Adults
Acronym: BCV-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EBS-BCV-001
Record Dates: First submitted 2023-06-05; First posted 2023-07-07 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Smallpox
Keywords: Smallpox; Pharmacokinetics (PK); Bioequivalence (BE); Orthopox; CMX001-129
MeSH Terms: conditions — Smallpox | interventions — brincidofovir

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-dose, randomized, two-period, crossover study to evaluate BE of BCV plasma PK parameters after administration of single 100 mg doses of BCV using the Form H (test tablet) and Form II (reference tablet) under fasting conditions in normal healthy adults. The study will also evaluate the safety of BCV following administration of two 100 mg single doses of BCV.
  Eligible participants will be randomized in a 1:1 ratio to one of two treatment sequences, Treatment AB or Treatment BA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment AB - Form H (test tablet) first (Active Comparator): Treatment AB:
  Participants assigned to Treatment AB in Period 1, will be given a single 100 mg tablet of Form H (test tablet). In Period 2, participants will be given a single 100 mg tablet of Form II (reference tablet) after a 14 day washout period.
  Interventions: Drug: Brincidofovir
- Treatment BA - Form II (reference tablet) first (Active Comparator): Treatment BA:
  Participants assigned to Treatment BA in Period 1, will be given a single 100 mg tablet of Form II (reference tablet). In Period 2, participants will be given a single 100 mg tablet of Form H (test tablet) after a 14 day washout period.
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — 100 mg tablet of Form H and 100 mg tablet of Form II
  Other Names: CMX001-129

SUMMARY:
The goal of this clinical trial is to evaluate whether both Form H and Form II, 100mg brincidofovir tablets are bioequivalent, when given under fasting conditions in healthy adults.

Participants will be randomized to each receive one tablet of Form H and one tablet of Form II,14 days apart and undergo pharmacokinetic testing pre-dose and post-dose to evaluate safety. This is an open-label, single-dose, randomized, two-period, crossover study.

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate the bioequivalence (BE) of brincidofovir (BCV) hydrate (Form H) tablet and the Form II tablet when administered under fasting conditions in healthy adult participants.
* To characterize plasma BCV pharmacokinetics (PK) following single doses of BCV when administered in healthy adult participants.

Safety Objective:

- To evaluate the safety of BCV following administration of single dose of 100 mg BCV Form H and BCV Form II tablet in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent voluntarily signed by participant.
* Male or female between 18 to 70 years of age, inclusive at screening.
* Body mass index (BMI) from 18 to 32 kg/m² with a minimum body weight of ≥ 50 kg, inclusive at screening.
* Women must be of nonchildbearing potential, i.e., postmenopausal woman (defined as spontaneous amenorrhea for 1-year prior to Period 1 Day 1) with a confirmed follicle stimulating hormone (FSH) level in laboratory's "postmenopausal" reference range; or a premenopausal woman documented as surgically sterile following either a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, tubal ligation.
* Males must be surgically sterilized (confirmed by documented azoospermia at least 90 days after procedure).
* Overtly healthy as determined by medical evaluation and judgment of the investigator including medical history, physical examination (PE), laboratory tests, vital signs (VS), and eletrocardiogram (ECG) at screening and Day -1. [Note: hematology, serum chemistry, and urinalysis parameters must fall within the laboratory's normal reference ranges or have been determined by the investigator to have no clinical significance in the context of this study.] Except:

  1. Alanine transaminase (ALT), aspartate aminotransferase (AST) and gammaglutamyl transferase (GGT) x ≤1.5 upper limit of normal reference range (ULN)
  2. Total Bilirubin x ≤1.5 ULN
  3. Hemoglobin (Hb) ≥10.5 g/dL for females or ≥12 g/dL for males
* Able to comply with the dosing instructions and available to complete the study schedule of assessments.

Exclusion Criteria:

* History or current symptoms of any serious psychiatric illness, including addiction, which could interfere with participant treatment, assessment, or compliance with the protocol.
* History of chronic liver disease or hepatic impairment, including but not limited to alcoholic liver disease, chronic viral hepatitis, autoimmune hepatitis, steatosis, or hemochromatosis. Note: A remote (≥12 months prior to screening) history of hepatitis A infection will not be cause for exclusion.
* History of Gilbert's syndrome or current evidence of the disease based on laboratory information at screening visit or Day -1.
* History of hematological disorders, including disorders such as a bleeding disorder or a risk of gastrointestinal bleeding.
* Clinically significant history of difficulty with blood donation, including vasovagal syncope (fainting), and/or poor venous access for the purposes of phlebotomy.
* Positive (reactive) serological test result at the screening evaluation consistent with possible infection with Hepatitis B virus (HBV), Hepatitis C virus (HCV), or Human immunodeficiency virus type 1 or 2 (HIV).
* Positive test for drugs of abuse and/or alcohol at either screening or check-in days.
* Clinically significant infection (e.g., COVID-19, cold, flu, or febrile illness) within 14 days prior to Period 1 Day 1.
* Donated a unit of blood or had clinically significant blood loss within 30 days prior to Period 1 Day 1 or donated plasma within 14 days prior to Period 1 Day 1.
* Received any investigational drug, agent, or device within 30 days prior to Period 1 Day 1, or current participation in another interventional study.
* Consumed any fruit juice including grapefruit juice, pomegranate juice, cranberry juice, orange juice, and Seville orange juice (also known as sour, bitter or bigarade orange) within 3 days prior to Period 1 Day 1 and throughout the study, unless prior approval is granted by both the investigator and the medical monitor.
* Received any medication or herbal product (e.g., St. John's wort) known to induce or inhibit hepatic metabolizing enzymes and/or transporters within 30 days or 5 half-lives of the compound, whichever is longer, prior to Period 1 Day 1 and throughout the study, unless approval is granted by both the investigator and the medical monitor.
* Received any vaccines (including COVID-19 vaccine) within 14 days prior to Period 1 Day 1 and throughout the study, unless approval is granted by both the investigator and the medical monitor.
* Any condition or set of circumstances that, in the judgment of the investigator, could interfere with the participant's ability to comply with the dosing schedule and completion of the study evaluations (e.g., participants who are unable to communicate or cooperate with the investigator).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
PK endpoint - Peak Plasma Concentration (Cmax) | Through 96 hours post-dose
  Assess maximum observed plasma concentration of Brincidofovir
PK endpoint - AUClast | Through 96 hours post-dose
  Assess area under the plasma concentration-time curve from time 0 to time of the last measurable concentration (AUC 0 - last) of Brincidofovir
PK endpoint - AUCinf | Through 96 hours post-dose
  Assess area under the plasma concentration-time curve from time 0 to infinity (AUC 0 - inf) of Brincidofovir
Incidence of treatment adverse events (AEs) | Through end of study visit (within 14 days after 2nd dose)
  Incidence of treatment-emergent AEs, treatment-related AEs, severe AEs, AEs leading to withdrawal and serious adverse events
Descriptive statistical summary abnormal Heart Rate | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of abnormal heart rate
Descriptive statistical summary abnormal Respiratory Rate | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of abnormal respiratory rate
Descriptive statistical summary abnormal Systolic Blood Pressure and Diastolic Blood Pressure (mmHg) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of abnormal Systolic Blood Pressure
Descriptive statistical summary abnormal Body Temperature (Celsius) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of abnormal body temperature
Chemistry parameters: Total Protein, Albumin, Globulin (g/dL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of Total Protein, Albumin, Globulin
Chemistry parameter: Albumin/Globulin ratio | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of albumin/globulin ratio
Chemistry parameters: alkaline phosphatase, ALT, AST, GGT and Creatine phosphokinase (U/L) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of alkaline phosphatase, ALT, AST, GGT and Creatine phosphokinase
Chemistry parameters: bilirubin (total and direct), BUN, serum calcium, glucose (random), serum phosphate, serum uric acid and serum magnesium (mg/dL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of bilirubin (total and direct), BUN, serum calcium, glucose (random), serum phosphate, serum uric acid and serum magnesium
Chemistry parameters: serum chloride, CO2, serum sodium and serum potassium (mmol/L) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of serum chloride, CO2, serum sodium and serum potassium
Chemistry parameter: Creatinine (g/24h) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of creatinine
Chemistry parameter: eGFR (ml/min) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of eGFR
Chemistry parameter: LDH (units/L) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of LDH
Hematology parameters: basophils, eosinophils, lymphocytes, monocytes and neutrophils (cells/uL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of basophils, eosinophils lymphocytes, monocytes and neutrophils
Hematology parameters: leukocytes and platelets (thousand/uL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of leukocytes and platelets
Hematology parameters: proportion of basophils, eosinophils, lymphocytes, monocytes and neutrophils | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of basophils/leukocytes, eosinophils//leukocytes, lymphocytes//leukocytes, monocytes//leukocytes and neutrophils//leukocytes
Hematology parameter: erythrocytes (million/uL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of erythrocytes
Hematology parameter: erythrocytes mean corpuscular volume (MCV) (fL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of erythrocytes MCV
Hematology parameter: hematocrit (%) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of hematocrit
Hematology parameter: hemoglobin (g/dL) | Through end of study visit (within 14 days after 2nd dose)
  Descriptive statistical summary (summarized by treatment, study day, and time) of hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Dave Cassie, MSc, Study Director — Director, Clinical Research
Locations (1):
- Altasciences, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No